CLINICAL TRIAL: NCT01026727
Title: A Phase 2b Multicenter, Randomized, Open Label, Comparative Trial of MPC-4326 in Combination With a Two to Three Drug Optimized Background Regimen Versus an Optimized, Three to Four Drug Antiretroviral Regimen for the Treatment of Triple Class Antiretroviral Experienced, HIV-1 Infected Subjects Failing Current Therapy
Brief Title: A Study to Assess the Long-term Efficacy (24 Weeks) of MPC-4326 in Combination With a 2-3 Drug OBR Relative to the Efficacy of a 3-4 Drug ARV Regimen in Treatment Experienced HIV-1 Infected Subjects Who Are Failing Current Antiretroviral Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For strategic buisness reasons.
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew Beelen, MD, Myriad Pharmaceuticals, Inc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-4326-003.01
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Virus Diseases; Sexually Transmitted Diseases, Viral; RNA Virus Infections; Slow Virus Diseases; Immune System Diseases; Sexually Transmitted Diseases; Lentivirus Infections; Infection; Retroviridae Infections; Immunologic Deficiency Syndromes; HIV; treatment experienced; bevirimat
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Virus Diseases; Sexually Transmitted Diseases, Viral; RNA Virus Infections; Slow Virus Diseases; Immune System Diseases; Sexually Transmitted Diseases; Lentivirus Infections; Infections; Retroviridae Infections; Immunologic Deficiency Syndromes | interventions — bevirimat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPC-4326 plus a 2-3 drug optimized background regimen (OBR) (Experimental): MPC-4326 300 mg or 400mg BID plus a 2-3 drug optimized background regimen (OBR)for 24 weeks.
  Interventions: Drug: MPC-4326 plus a 2-3 drug optimized background regimen (OBR)
- 3-4 drug antiretroviral drugs (Active Comparator): 3-4 commercially available antiretroviral (ARV)drugs for 24 weeks.
  Interventions: Drug: 3-4 commercially available antiretroviral drugs

INTERVENTIONS:
Drug: MPC-4326 plus a 2-3 drug optimized background regimen (OBR) — For treatment arm #1: the MPC-4326 dose will be selected based on the inclusion of raltegravir (i.e., will be limited to 300 mg BID) or inclusion of darunavir (i.e., will be assigned 400 mg BID) in the OBR. If both raltegravir and darunavir are included in the OBR for a subject, the subject will be limited to 300 mg BID
  Arms: MPC-4326 plus a 2-3 drug optimized background regimen (OBR)
Drug: 3-4 commercially available antiretroviral drugs — For treatment arm #2: the antiretroviral regimen, dosage and frequency will be selected by the investigator.
  Arms: 3-4 drug antiretroviral drugs

SUMMARY:
This phase 2b study is designed to assess the long-term efficacy (24 weeks) of MPC-4326 in combination with a 2-3 drug optimized background regimen (OBR) relative to the efficacy of a 3-4 antiretroviral (ARV) regimen in treatment experienced, HIV-1 infected subjects.

DETAILED DESCRIPTION:
Standard antiretroviral therapies for the treatment of HIV/AIDS, while effective for varying lengths of time, can be rendered inadequate for viral suppression by the emergence of drug resistant virus, which can include resistance to entire mechanistic classes of drugs. Thus, there exists a significant unmet medical need for new highly potent antiretroviral agents with novel mechanisms of action. The novel mechanism of action of MPC-4326 suggests that MPC-4326 may have utility for the treatment of HIV-1 infected patients failing current regimens due to the development of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consent to participate in the study (sign Informed Consent Form), and able to understand study procedures and complete the study.
2. Be at least 18 years of age at the time of screening.
3. Have a screening plasma HIV-1 RNA value ≥ 1,000 copies/mL
4. Be receiving an ARV regimen containing at least 3 drugs which has been unchanged for at least 8 weeks prior to initial screening.
5. Have at least two fully active ARVs (exclusive of MPC-4326) as determined by a 'maximal response' on the vircoTYPE assay; R5 tropism testing (if applicable); and treatment history (e.g., naïve to enfuvirtide or integrase inhibitors) that can be combined in a regimen containing a maximum of four ARVs for the 3-4d ARV regimen or three ARVs for the 2-3-drug OBR to be combined with MPC-4326.
6. Two NRTIs are not allowed as the only fully-active antiretroviral agents in the 3-4-drug ARV regimen or in the 2-3-drug OBR
7. Must have wild type Gag at position 370 (i.e., no polymorphisms at 370)
8. Have resistance to at least one agent in each of the three 'classic' ARV drug classes (NRTI, NNRTI, PI) to include documented evidence of resistance on prior resistance tests.
9. Females of childbearing potential must agree to the use two forms of contraception from the time of screening until 90 days after completion of dosing.Surfactant-type spermicide gels and contraceptive foam are not recommended, as they increase the rate of HIV transmission.

Exclusion Criteria:

1. Be pregnant or breast feeding
2. Presence of any significant acute illness (as determined by the investigator) within 14 days of study entry.
3. Presence of any AIDS-related opportunistic infection (Category C according to the CDC Classification System for HIV-1 Infection, 1993 Revised Version) that is unstable in the Investigator's opinion or diagnosed in the 30 days prior to study entry (i.e., Run in Period Day 1).
4. A history of cerebrovascular accident or transient ischemic attacks.
5. Subjects with the following laboratory parameters within 14 days prior to first dose of study drug:

   1. Hemoglobin < 10 g/dL for men and < 9 g/dL for women
   2. Absolute neutrophil count < 1000/mm3
   3. Platelet count < 50,000/mm3
   4. AST or ALT > 5 times the upper limit of normal inclusive of subjects with a positive HBV surface antigen or HCV antibody test at screening
   5. Calculated creatinine clearance (ClCr) <40 mL/min as determined by the Cockcroft-Gault equation
6. Subjects who have received radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to the first dose of study drug.
7. Subjects who have received treatment with immunomodulating agents such as IL-2, α IFN, β IFN or γ IFN within 4 weeks prior to the first dose of study drug.
8. Subjects who use or require a prohibited therapy within 30 days prior to or while participating in this study.
9. Receipt of an investigational drug or product, or participation in a drug study within a period of 30 days prior to receiving study medication. For investigational drugs with an elimination half life greater than 10 days, this period will be extended to 60 days and for antibody-based products (i.e., CD4 antibody products, etc.) this period will be extended to 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a viral load <50 copies/mL at 24 weeks in each treatment group | 24-weeks

SECONDARY OUTCOMES:
The key secondary endpoint is to compare the Viral Load Decrease at 24 weeks in the two treatment arms. VLD is defined as the change from baseline log10 viral load. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.
Locations (25):
- United States (21):
  - AIDS Healthcare Foundation Research Center, Beverly Hills, California
  - Peter Wolfe, MD, PC, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond, MD, PA, Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Community Research Initiative of New England, Boston, Massachusetts
  - University of Rochester , Strong Memorial Hospital, Rochester, New York
  - North Bronx Health Care Network, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Kaiser Permanente Immune Deficiency Clinic, Portland, Oregon
  - Central Texas Clinical Research, Austin, Texas
  - Southwest Infectious Disease, Dallas, Texas
  - North Texas Infectious Disease Consultants, PA, Dallas, Texas
  - Therapeutic Concepts, P.A, Houston, Texas
  - DCOL Center, Longview, Texas
  - CARE-ID, Annandale, Virginia
  - EHS Pulmonary & Critical Care, Spokane, Washington
- Canada (4):
  - University of British Columbia,Downtown Infectuous Diseases Clinic, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique médicale l'Actuel,, Montreal, Quebec
  - Clinique Médicale Quartier Latin, Montreal, Quebec